CLINICAL TRIAL: NCT06372600
Title: Effect of Extracorporeal Shock Wave Combined With Autologous Platelet-rich Plasma Injection on Rotator Cuff Calcific Tendinitis: A Randomized Controlled Trial
Brief Title: Effect of Extracorporeal Shock Wave Combined With Autologous Platelet-rich Plasma Injection on Rotator Cuff Calcific Tendinitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiali Xue (Other)
Responsible Party: Sponsor-Investigator, Xiali Xue, Clinical Professor, Chengdu Sport University
Organization: Chengdu Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-181
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tendinitis; Rotator Cuff Tendinosis
Keywords: Rotator cuff calcifying tendinitis; PRP; ESW
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extracorporeal shock wave therapy group (Experimental): In the shoulder pain points, choose 2 to 3 of them for each treatment, apply the coupling agent, which is convenient for the treatment head to stick to the skin, and complete the longitudinal treatment and horizontal treatment. The setting frequency was 4 ~ 8 Hz, the length of the probe was 15 mm, and the pressure was set at 1.5 mJ/mm2. The frequency of each treatment point reached 2 000 ~ 2 500 times, and the hand-held pressure was set to medium-high level. A total of 6 treatments were completed. For patients with unclear pain points or regional pain, the treatment point should be supraspinatus tendon or infraspinatus tendon, and the treatment should be completed with the most severe pain site.
  Interventions: Device: Extracorporeal shock wave therapy device
- Platelet-rich plasma group (Experimental): Autologous Platelet-rich plasma injection was performed under ultrasound guidance
  Interventions: Biological: Platelet-rich plasma
- Extracorporeal shock wave therapy+Platelet-rich plasma group (Experimental): Extracorporeal shock wave therapy followed by Platelet-rich plasma injection
  Interventions: Device: Extracorporeal shock wave therapy device; Biological: Platelet-rich plasma

INTERVENTIONS:
Device: Extracorporeal shock wave therapy device — In the shoulder pain points, choose 2 to 3 of them for each treatment, apply the coupling agent, which is convenient for the treatment head to stick to the skin, and complete the longitudinal treatment and horizontal treatment. The setting frequency was 4 ~ 8 Hz, the length of the probe was 15 mm, and the pressure was set at 1.5 mJ/mm2. The frequency of each treatment point reached 2 000 ~ 2 500 times, and the hand-held pressure was set to medium-high level. A total of 6 treatments were completed. For patients with unclear pain points or regional pain, the treatment point should be supraspinatus tendon or infraspinatus tendon, and the treatment should be completed with the most severe pain site.
  Arms: Extracorporeal shock wave therapy group; Extracorporeal shock wave therapy+Platelet-rich plasma group
Biological: Platelet-rich plasma — Autologous Platelet-rich plasma injection was performed under ultrasound guidance
  Arms: Extracorporeal shock wave therapy+Platelet-rich plasma group; Platelet-rich plasma group

SUMMARY:
The purpose of this study is to explore the effect of extracorporeal shock wave combined with autologous platelet-rich plasma injection on the rehabilitation of rotator cuff calcific tendinitis, to provide new treatment methods and evidence for the rehabilitation of rotator cuff calcific tendinitis, and to reduce patients; pain and return to normal life as soon as possible.

DETAILED DESCRIPTION:
The purpose of this study is to explore the effect of extracorporeal shock wave combined with autologous platelet-rich plasma injection on the rehabilitation of rotator cuff calcific tendinitis, to provide new treatment methods and evidence for the rehabilitation of rotator cuff calcific tendinitis, and to reduce patients' pain and return to normal life as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for rotator cuff calcific tendonitis, aged between 40 and 60 years old
* Persistent pain in the affected shoulder, with obvious tenderness under the acromion and rotator cuff, as confirmed by X-ray and Computed Tomography (CT) and Magnetic Resonance Imaging (MRI) examination showed one or more round-shaped high-density calcium salt deposits near the greater tuberosity of the humerus
* All were diagnosed for the first time
* Complaints of severe pain in the shoulder joint, obvious

Exclusion Criteria:

* Combined with rotator cuff trauma, long head of biceps tendonitis and other shoulder joint diseases
* Past combined history of shoulder joint surgery
* Patients with internal fixation of the shoulder joint
* Shoulder joint combined with infection, Tumors and other lesions
* Combined with severe heart, liver, and kidney dysfunction
* Do not agree to participate in the study or fail to sign the informed consent form.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale,VAS | After 1, 2, 4 and 8 weeks of intervention
  The full name of the Scale is Visual Analogue Scale, that is, visual analogue scale.
  Minimum value and maximum value: the minimum value of the VAS scale is 0, indicating "completely painless" or "painless end"; The maximum value is 10, which indicates "the most severe pain imaginable" or "the most severe pain end." Score Significance: On the VAS scale, a higher score means a worse outcome, i.e. a greater degree of pain. The patient marks the corresponding position on the scale according to their pain experience, thus indicating the intensity of the pain.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeon's Form,ASES | After 1, 2, 4 and 8 weeks of intervention
  The full name of the scale: American Shoulder and Elbow Surgeons Score, namely, American Shoulder and Elbow Surgeons Score.
  Minimum value and maximum value: The minimum value of ASES scale is 0 and the maximum value is 100.
  Score Significance: On the ASES scale, a higher score means a better outcome, i.e. a better functional state of the shoulder or a milder condition.
the university of California at Los Angeles shoulder rating scale, UCLA | After 1, 2, 4 and 8 weeks of intervention
  Full name of the Scale: University of California at Los Angeles Shoulder Rating Scale.
  Minimum and maximum values: The minimum value of the UCLA Shoulder Joint Scoring Scale is usually 0, and the maximum value may vary depending on the version and scoring rules, but a common maximum value is 35.
  Score Significance: On the UCLA Shoulder Joint Rating Scale, a higher score generally means a better outcome, i.e. better shoulder function or less pain.
The location and size of the calcifications were examined by ultrasound | After 4 and 8 weeks of intervention

IPD SHARING:
Plan to Share IPD: No
To protect patient privacy, the investigators have chosen not to share data for the time being.

REFERENCES:
- [Derived] Wang X, Jia S, Cui J, Xue X, Tian Z. Effect of extracorporeal shock wave combined with autologous platelet-rich plasma injection on rotator cuff calcific tendinitis: study protocol for a randomized controlled trial. Trials. 2024 Sep 18;25(1):616. doi: 10.1186/s13063-024-08407-z. PMID 39294797